CLINICAL TRIAL: NCT03864575
Title: NICE-COMBO: An Open Label Phase II Study Combining Nivolumab and Celecoxib in Patients With Advanced " Cold " Solid Tumors
Brief Title: An Open Label Phase II Study Combining Nivolumab and Celecoxib in Patients With Advanced " Cold " Solid Tumors
Acronym: NICE-COMBO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUC-19-002
Record Dates: First submitted 2019-02-28; First posted 2019-03-06 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Cancer
Keywords: Nivolumab; Celecoxib
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Celecoxib; Nivolumab

STUDY DESIGN:
Intervention Model Description: Simon's two-stage Minimax design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination Group (Experimental): Celecoxib 400 mg/d Nivolumab 240 mg q2w
  Interventions: Drug: Celecoxib 400 mg

INTERVENTIONS:
Drug: Celecoxib 400 mg — Celecoxib 400 mg/day in combination with nivolumab fixed dose
  Other Names: Nivolumab 240 mg q2w

SUMMARY:
This is an open-label study to evaluate the safety and the anti-tumor activity of the combination of nivolumab and celecoxib.

The total numbers of participants to be enrolled will be up to 68 participants, depending on the investigated dose of celecoxib during the safety run-in phase.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Measurable disease as per RECIST 1.1.
* Adequate renal, hepatic and hematologic functions as defined by laboratory parameters within ≤ 7 days before treatment initiation.
* Metastases biopsiable on two occasions
* Recently acquired (within 90 days prior to treatment) tumor tissue from an unresectable or metastatic site of disease must be provided for biomarker analyses. In order to include only IDO1 positive (≥5% expression of tumor cells) and non T-cell infiltrated tumors (<1% T cells infiltrating the tumor bed)
* Cancer types with an indication of treatment with anti-PD1 antibodies such as

  * Melanoma non BRAF mutated in first line of treatment
  * Melanoma BRAF mutated in first or second line of treatment
  * Lung cancer (NSCLC) in second line of treatment
  * Renal cell Cancer (RCC) in second line of treatment
  * Head and Neck squamous carcinoma (HNSC) after platinum salt based chemotherapy
  * Bladder cancer after platinum salt based chemotherapy

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases.
* Ocular melanoma.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement therapy, psoriasis not requiring systemic treatment, or other autoimmune condition not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects must also meet other study criteria including exclusions for medical history, positive Hep B/C, HIV, and pregnancy tests, and other laboratory criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-08-15 (Estimated); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
objective response rate | at week 12 from onset of treatment
  To evaluate the objective response rate (ORR) of Celecoxib in combination with anti-PD1 antibodies

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | from first dose to day 28 post last dose
  All the patients that will receive at least one dose of nivolumab and celecoxib are assess for toxicity endpoint. All adverse events will be recorded and graded based on the CTCAE v4.0 scale.
  antibodies
Efficacy - Duration of response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  defined as the time from earliest date of CR or PR (as determined by investigator assessment of radiographic disease burden per RECIST v1.1) until the earliest date of disease progression or death, due to any cause, if occurring sooner than disease progression.
Efficacy - Time to response (TTR) | From onset of treatment to response of cancer through study completion, an average of 12 months is expected
  defined as the time from the date of first dose of study drug until the time of the earliest date of CR or PR (as determined by investigator assessment of radiographic disease burden per RECIST v1.1.
Disease control rate (DCR) | at week 12 from onset of treatment
  defined as the percentage of subjects having CR, PR, or stable disease (SD) for at least 8 weeks, as determined by investigator assessment of radiographic disease as per RECIST v1.1.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death, whichever comes first, assessed up to 60 months
  defined as the time from the date of first dose of study drug until the earliest date of disease progression (as determined by investigator assessment of radiographic disease burden per RECIST v1.1), or death due to any cause, if occurring sooner than progression.
Overall survival (OS) | From date of randomization until the date of death, assessed up to 60 months
  defined as the time from the date of first dose of study drug until death, due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Françoi Baurain, MD,PHD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Sain-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No